CLINICAL TRIAL: NCT01915004
Title: Bladder Training Video Versus Individual Urotherapy for Children With Non-neurogenic Lower Urinary Tract Dysfunction.
Brief Title: The Effectiveness of a Bladder Training Video for Management of Lower Urinary Tract Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Urological Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bladder Training Video
Record Dates: First submitted 2013-07-26; First posted 2013-08-02 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2017-08

CONDITIONS: Nonneurogenic Lower Urinary Tract Dysfunction; Dysfunctional Elimination Syndrome
Keywords: Pediatric Urology; Urotherapy; Nonneurogenic Lower Urinary Tract Dysfunction; Dysfunctional Elimination Syndrome; Randomized Controlled Trial
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Invididual Urotherapy (Other): Educational Intervention. Standard individual urotherapy (bladder re-training) occurs in the pediatric urology clinic.
  Interventions: Other: Educational Intervention
- Bladder Training Video (Experimental): Experimental Educational Intervention. Participants will watch a 7 minute animated bladder training video.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Bladder Training Video

SUMMARY:
Children with non-neurogenic lower urinary tract dysfunction (NLUTD) represent a significant subgroup of pediatric urology patients, comprising up to 30 percent of some out-patient clinics. These children present with urinary tract infections (UTIs), abnormal voiding habits and various other lower urinary tract symptoms (LUTs) such as incontinence, urinary urgency and urinary frequency. Furthermore, the effects of NLUTD on a child's physical health, mental health and its potential negative clinical sequelae, which includes upper or lower urinary tract damage, must be taken into account when treating these children. These patients have complex needs requiring a significant amount of health teaching and it is imperative to determine the effectiveness of the various modes of delivering urotherapy. To determine the best modality to deliver urotherapy, this trial will compare the effectiveness of a 7 minute bladder training video to the effectiveness of standard urotherapy provided at a pediatric urology clinic at improving NLUTD/DES symptoms and quality of life in children between 5-10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-10 years old
* Bladder Dysfunction (Diagnosis of NLUTD or DES)

Exclusion Criteria:

* Grade 3 or 4 hydronephrosis
* Grade 3, 4 or 5 vesicoureteral reflux
* Other diagnoses which affect bladder bowel function (i.e. Spina Bifida)
* English as a second language
* Diagnosed learning disability (i.e. ADD or ADHD)
* Mental health condition (i.e. anxiety or depression)
* Received intensive urotherapy and biofeedback in past 12 months
* Child is diagnosed with primary nocturnal enuresis

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Improvement of Nonneurogenic Lower Urinary Tract Dysfunction symptoms | up to 12 weeks
  Determine improvement of Nonneurogenic Lower Urinary Tract Dysfunction symptoms according to the Vancouver NLUTD/DES questionnaire after administration of either intervention (Bladder Training Video or standard urotherapy)

SECONDARY OUTCOMES:
Assess the Quality of Life of children with Nonneurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome. | Up to 12 weeks
  The secondary outcome is to assess the QOL of children with NLUTD/DES. QOL will be measured by a validated QOL tool specific to children with bladder dysfunction called the PinQ

CONTACTS AND LOCATIONS:
Overall Officials: Luis Braga, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada